CLINICAL TRIAL: NCT02323815
Title: The Effect of Integrated Prevention and Treatment on Child Malnutrition and Health in Mali: a Cluster Randomized Intervention Study
Acronym: PROMIS-Mali
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: Helen Keller International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IFPRI
Record Dates: First submitted 2014-12-18; First posted 2014-12-24 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Child Acute Malnutrition
Keywords: child acute malnutrition prevention; behavior change communication; lipid-based nutrient supplement; screening coverage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Behavior change communication (BCC) on Essential Nutrition Actions (ENA), Infant and Young Child Feeding (IYCF) and Water, sanitation and hygiene (WASH) is provided during monthly meetings for children 6-23 months of age
  Interventions: Behavioral: Child's health and nutrition topics
- PROMIS intervention (Experimental): * Behavior change communication (BCC) on Essential Nutrition Actions (ENA), Infant and Young Child Feeding (IYCF) and Water, sanitation and hygiene (WASH) is provided during monthly meetings for children 6-23 months of age
  * Caregivers with children 6-23 months of age that attend Counselling meetings will be provided with a monthly dose of SQ-LNS (20g/day)
  Interventions: Dietary Supplement: Small-Quantity Lipid-based nutrient supplement; Behavioral: Child's health and nutrition topics

INTERVENTIONS:
Dietary Supplement: Small-Quantity Lipid-based nutrient supplement — A monthly dose of SQ-LNS (31 sachets of 20g) will be distributed to mothers attending counselling sessions
  Other Names: SQ-LNS
  Arms: PROMIS intervention
Behavioral: Child's health and nutrition topics — Monthly group counselling meetings organized at village level. Caregivers of participating children are invited to attend monthly counselling meetings that treat topics on child nutrition, health, hygiene and good sanitary practices. During these visits children are also screened for acute malnutrition measuring arm circumference.

SUMMARY:
Globally, child undernutrition is the underlying cause for 3.1 million deaths of children younger than 5 years. 18.7 million children under five years of age suffer from severe acute malnutrition (SAM) and an additional 33 million children suffer from moderate acute malnutrition, and are at risk of developing SAM

In Sub-Saharan Africa, there is often poor integration between programs to treat child acute malnutrition and programs that focus on the prevention of acute and chronic undernutrition - resulting in many missed opportunities for using prevention platforms to screen and refer SAM children, or for using screening and referral platforms to provide prevention services.

This project will address two critical gaps related to the integration of preventive and treatment programs: 1) screening and treatment of MAM/SAM have not yet been systematically integrated into routine health-center visits or mainstreamed into community outreach programs; and 2) screening programs do not offer any preventive services for those children found not to be suffering from MAM/SAM at the time of screening; mothers of children identified as non-MAM/SAM case are usually sent home without receiving any health or nutrition inputs and as a result, may fail to come back for screening because they do not see any tangible benefit associated with their participation in the screening. This project will specifically address these gaps by assessing the effect of an integrated approach consisting of higher screening coverage and preventive Behavior Change Communication (BCC) + Small-Quantity Lipid-based Nutrient supplementation (SQ-LNS) on both prevention and treatment of child undernutrition.

DETAILED DESCRIPTION:
Because of the intended dual role of BCC/SQ-LNS on child undernutrition in this study - e.g. to help prevent child undernutrition and enhance the coverage of screening, referral and treatment of SAM/MAM, it is necessary to combine two study designs to rigorously evaluate the impact of the proposed intervention and to tease out the contribution of prevention and enhanced coverage/treatment to the overall impact on child malnutrition.

The proposed study will therefore use two types of study designs. The first one is a repeated cross-sectional design that will compare select study outcomes between intervention and control groups at endline, after 24 months of program implementation. These cross-sectional surveys among children 6-23 months, at baseline and after 24 months (on different children) will be used to assess the impact of the intervention on the prevalence of several outcomes, including the prevalence of MAM/SAM and stunting, the coverage of MAM/SAM screening and maternal ENA/IYCF/WASH knowledge and practices. The second study design entails a longitudinal design whereby individual children will be recruited at 6 months of age and followed-up monthly until they reach 24 months of age.This design will allow us to assess the intervention's effects on the incidence, recovery and recurrence rates of MAM/SAM.

ELIGIBILITY:
Cross-sectional study (baseline and endline)

Inclusion Criteria:

* At least one index child 6-23 months of age in the household
* Mother should be living in the study area since the index child's delivery
* Singleton infants

Exclusion Criteria:

* Index child should not present congenital deformations that hamper anthropometric measurements

Longitudinal study

Inclusion Criteria:

* Child 6-6.9 months of age;
* Child with WHZ>-2 and MUAC>125 mm and no bilateral pitting edema
* Mother should be living in the study area since the index child's delivery
* Singleton infants

Exclusion Criteria:

* Congenital malformations that make anthropometric measurements impossible
* Mother planning to leave the study are in the coming year

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2304 (Estimated)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of acute child malnutrition defined by WHZ<-2 or MUAC <125mm or bilateral pitting edema in children 6-23 months of age | After 24 months of program implementation
  * Cross-sectional study
  * To calculate WHZ scores the 2006 WHO growth reference will be used
Screening coverage of acute child malnutrition (proportion of children monthly screened / total number of eligible children (aged 6-23 months) | monthly from study inclusion at 6 months to 23 months of age and at study endline
  * Cross-sectional study
  * Longitudinal study
Incidence of child acute malnutrition defined by WHZ<-2 or MUAC<125mm | Monthly from study inclusion at 6 months to 23 months of age
  * Longitudinal study
  * To calculate WHZ scores the 2006 WHO growth reference will be used
Compliance to treatment of acute malnutrition (% of cases that complete treatment over total admitted) | monthly from study inclusion at 6 months to 23 months of age and at study endline
  * Cross-sectional study
  * Longitudinal study

SECONDARY OUTCOMES:
Prevalence of child stunting defined by HAZ<-2 in children 6-23 months of age | After 24 months of program implementation
  To calculate HAZ scores the 2006 WHO growth reference will be used
Mean WHZ-score in children 6-23 months of age | After 24 months of program implementation
  To calculate WHZ scores the 2006 WHO growth reference will be used
Mean HAZ-score in children 6-23 months of age | After 24 months of program implementation
  To calculate HAZ scores the 2006 WHO growth reference will be used
Mean Mid-Upper Arm Circumference in children 6-23 months of age | After 24 months of program implementation
Mean hemoglobin concentration at endline in children 6-23 months of age | After 24 months of program implementation
Prevalence of child anemia (Hb concentration<11g.dL-1) at endline in children 6-23 months of age | After 24 months of program implementation
Prevalence of Severe Acute Malnutrition defined by a WHZ<-3 or bilateral pitting edema or a MUAC<115mm | After 24 months of program implementation
  To calculate WHZ scores the 2006 WHO growth reference will be used
Prevalence of severe stunting defined by a HAZ<-3 in children 6-23 months of age | After 24 months of program implementation
  To calculate HAZ scores the 2006 WHO growth reference will be used
Caregiver's knowledge and practices related to Infant and Young Child Feeding (IYCF), Essential Nutrition Actions (ENA) and Water, Sanitation and Hygiene (WASH) | After 24 months of program implementation
Incidence of child stunting defined by HAZ<-2 in children from 6 to 23 months of age | monthly from inclusion at 6 months to 23 months of age
  To calculate HAZ scores the 2006 WHO growth reference will be used
Linear growth velocity (HAZ increment/month) | monthly from inclusion at 6 months to 23 months
  To calculate HAZ scores the 2006 WHO growth reference will be used
Ponderal growth velocity (WHZ increment/month) | monthly from inclusion at 6 months to 23 months
  To calculate WHZ scores the 2006 WHO growth reference will be used
Weight gain (weight increment/month) | monthly from inclusion at 6 months to 23 months
Mid-Upper Arm Circumference gain (MUAC increment /month) | monthly from inclusion at 6 months to 23 months
Infant morbidity (acute respiratory infections, fever, malaria (RDT), vomiting, diarrhea) | monthly from inclusion at 6 months to 23 months
  Malaria will be tested in case of fever (or recalled fever over last 24 hrs) using rapid tests
Relapse rate after treatment of MAM/SAM (proportion WHZ<-2 or MUAC<125mm or bilateral pitting edema after discharge from MAM or SAM treatment program over a total number of children treated | monthly from inclusion at 6 months to 23 months
Child development (motor, language and personal-social development) | After 24 months of program implementation
  Determined by DMC-II

CONTACTS AND LOCATIONS:
Overall Officials: Marie Ruel, PhD, Study Director — International Food Policy Research Institute; Harouna Konde, MD, Principal Investigator — Helen Keller International - Mali; Lieven Huybregts, PhD, Principal Investigator — International Food Policy Research Institute; Agnes Le Port, Principal Investigator — International Food Policy Research Institute
Locations (1):
- Bla and San Health Districts, Bla and San, Ségou, Mali

REFERENCES:
- [Derived] Huybregts L, Le Port A, Becquey E, Zongrone A, Barba FM, Rawat R, Leroy JL, Ruel MT. Impact on child acute malnutrition of integrating small-quantity lipid-based nutrient supplements into community-level screening for acute malnutrition: A cluster-randomized controlled trial in Mali. PLoS Med. 2019 Aug 27;16(8):e1002892. doi: 10.1371/journal.pmed.1002892. eCollection 2019 Aug. PMID 31454356
- [Derived] Huybregts L, Becquey E, Zongrone A, Le Port A, Khassanova R, Coulibaly L, Leroy JL, Rawat R, Ruel MT. The impact of integrated prevention and treatment on child malnutrition and health: the PROMIS project, a randomized control trial in Burkina Faso and Mali. BMC Public Health. 2017 Mar 9;17(1):237. doi: 10.1186/s12889-017-4146-6. PMID 28274214